CLINICAL TRIAL: NCT00146913
Title: A Phase II Study Evaluating the Efficacy and Tolerance of Combination Therapy of Imatinib Mesylate (IM) +-2A Interféron for Chronic Phase CML Patients Resistant or Refractory to IM Used as Single Therapy for at Least One Year
Brief Title: AFR10 - Combination Therapy of Imatinib Mesylate (IM) + Alpha-2A Interferon for Chronic Phase CML Patients Resistant or Refractory to IM Used as Single Therapy for at Least One Year
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Hospices Civils de Lyon (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: 2003.317
Record Dates: First submitted 2005-09-05; First posted 2005-09-07 (Estimated); Last update posted 2007-04-27 (Estimated); Status verified 2007-04

CONDITIONS: Chronic Myeloid Leukemia
Keywords: Chronic myeloid leukaemia; resistant; refractory; Imatinib mesylate
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive | interventions — Imatinib Mesylate

INTERVENTIONS:
Drug: Imatinib mesylate 600mg/day
Drug: Peg-Interféron at 90 microg/week

SUMMARY:
Sixty % of CML patients treated by Imatinib mesylate achieved a major cytogenetic responses (CCR) at 18 months. So, 40% of the patients must receive additional treatment. In vitro, it has been shown that IM and Interféron-alpha have synergic anti-proliferative effect on chromosome Ph+ cell lines. By using Peg-Interféron and IM combination, we hope to increase the cytogenetic response of patients.

ELIGIBILITY:
Inclusion Criteria:

* Chronic phase Philadelphia positive CML, confirmed by karyotyping (or FISH) analysis, in complete hematologic response with IM.
* Lack of major cytogenetic response after at least one year of STI 571 as single therapy.
* Male and female * 18 years old.
* Informed consent signed up.
* Performance status grade 0 - 2 (ECOG).
* SGOT and SGPT <3N
* Serum bilirubin < 1.5 N
* Serum creatinine < 1.5 N
* No HSC graft planned
* B-HCG negative for female with potential childbearing

Exclusion Criteria:

* Absence of complete hematologic response
* Extramedullar involvement
* Previous extra-hematologic intolerance of Interféron at a dose superior or equal to 25 MUI/week
* Depressive syndrome not controlled
* Not controlled dysthyroidy
* Auto-immune pathology not controlled
* Women with childbearing potential who are unwilling or unable to use an adequate method to avoid pregnancy for the entire period of the study
* Significant cardiac disease (grade 3 or more)
* Known seropositivity for HIV
* Active viral hepatitis
* Other malignant disease
* Other experimental medication

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30
Dates: Start 2004-03

PRIMARY OUTCOMES:
Study the maintenance of a complete hematologic response, the cytogenetic and molecular responses, and the overall survival of the patients population

SECONDARY OUTCOMES:
Evaluate the tolerance of a combination of STI571 and alpha-interferon

CONTACTS AND LOCATIONS:
Overall Officials: Mauricette MICHALLET, MD, Principal Investigator — Hospices Civils de Lyon
Locations (1):
- Franck NICOLINI, Lyon, France